CLINICAL TRIAL: NCT02695433
Title: Effects of a Typical American Diet High in Refined Carbohydrates Compared to a Diet That Replaces Some Refined Carbohydrates With Healthy Fats on Cardiometabolic Health in Men and Women With Pre-diabetes and Metabolic Syndrome
Brief Title: Replacing Refined Carbohydrates With Healthy Fats on Cardio-metabolic Markers
Acronym: AV2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB2016-001
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Pre-diabetes; Metabolic Syndrome
Keywords: Pre-diabetes; Metabolic syndrome; Matsuda composite index of insulin sensitivity (MISI); Blood glucose; Insulin response; HbA1c; Lipid; Inflammation
MeSH Terms: conditions — Glucose Intolerance; Metabolic Syndrome; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment (AT) diet plan (Experimental): 1 Avocado 7 days/week (5-7 days is acceptable) over a 12 week period
  Interventions: Dietary Supplement: Active
- Control (CT) diet plan (Placebo Comparator): at least 1 serving of a low fat, low fiber, high glycemic carbohydrate and eliminate avocado 7 days / week (5-7 days is acceptable) over a 12 week period
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Active — Active Treatment Diet Plan
  Arms: Active treatment (AT) diet plan
Dietary Supplement: Control — Control Diet Plan
  Arms: Control (CT) diet plan

SUMMARY:
The primary goal is to to characterize the effects of consuming 1 avocado fruit 7 days / week (5-7 days is acceptable) compared to a no avocado relatively low fat, carbohydrate control treatment over a 12 week period on insulin sensitivity as measured by the Matsuda composite index of insulin sensitivity (MISI).

DETAILED DESCRIPTION:
The trial is designed as a randomized, controlled, statistician blinded, 2-arm parallel study to investigate the effects of avocado consumption compared to non-avocado control foods which have opposing macronutrients (avocado is relatively higher in fat and in low carbohydrate and the control foods will be low fat, high carbohydrate options) on indices of cardiometabolic health over a 12 week period.

The trial will test 2 treatment conditions in pre-diabetic men and women 25-60 years of age with metabolic syndrome. One hundred twenty men and women will be recruited, aiming for a completer set of 96 subjects. Qualified Subjects will be randomized to receive 1 of 2 test treatments based on randomization schedule from a computer generated randomization schedule.

Study treatments include:

* Control (CT) diet plan with at least 1 serving of a low fat, low fiber, high glycemic carbohydrate and eliminate avocado 7 days / week (5-7 days is acceptable) over a 12 week period.
* Active treatment (AT) diet plan will include 1 Avocado 7 days/week (5-7 days is acceptable) over a 12 week period.

Each subject will be asked to come for one Screening Visit, 9 interim food pick-up/compliance visits and 4 Test Day Visits. The four main Test Day visits will occur at week 0 (day 1; baseline), end of week 4, at the end of week 8 and at the end of week 12. Interim Visits will occur at week 1, 2, 3, 5, 6, 7, 9, 10 and 11. Subjects will pick-up study foods, answer questionnaires, receive dietary counseling, confirm diet compliance during interim visits. They will also be asked to complete online 24 hour food recalls up to once per each week of the study. Each of the 4 Test Day Visits will last about 2-3.5 h and involve blood pressure (BP) measurements, a fasting blood sample collection and anthropometric, body composition assessment. In addition, an oral glucose tolerance test (OGTT) will be performed at week 0/day 1 and at the end of week 12/day.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 25-65 yrs.
* BMI of 25 - 42 kg/m2
* HOMA-IR ≥ 2
* Abdominal obesity: mid-point waist circumference >102 cm for men and >88 cm for women
* No clinical evidence / history of heart disease, respiratory, renal, gastrointestinal, or hepatic disease
* Not taking over-the-counter or prescription medications/dietary supplements that may interfere with study procedures or endpoints (e.g., antioxidant supplements, protein powder, energy drinks, anti-inflammatory or lipid-lowering medications).
* Non-smoker or past smoker (smoking cessation > 2 yrs.)
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Aged < 25 or > 65 years
* BMI < 25 kg/m2 or > 42 kg/m2
* HOMA-IR < 2.0
* History of heart disease, respiratory, renal, gastrointestinal or hepatic disease
* Diabetes
* Have or had cancer other than non-melanoma skin cancer in past 5 years
* Taking over-the-counter or prescription medications or dietary supplements that may interfere with study procedures or endpoints (including protein powers, energy drinks)
* Vegan dietary habits, unusual dietary habits or sensitive or allergic to any of the test meal components / ingredients
* Consuming 3 or more avocados per week.
* Consuming 3 or more servings of nuts or peanuts per week, unless subject is willing to stop consuming nuts 4 weeks before and throughout the course of the study.
* Excessive coffee and tea consumers (>4 cups/day)
* Current smoker
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in 3 months
* Drug or alcohol addiction
* Present with significant psychiatric or neurological disturbances
* Working overnight (e.g 3rd shift of overnight workers)
* Pregnant, lactating or planning to become pregnant
* Have donated blood within 3 months of the screening visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Women who are taking unstable dose and brand of hormonal contraceptive and/or stable dose and brand less than 6 months
* Excessive exercisers or trained athletes
* Take part in chronic feeding or medication clinical trial in the last 3 months

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in insulin sensitivity as measured by the Matsuda composite index of insulin sensitivity (MISI) in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  insulin sensitivity as measured by the Matsuda composite index

SECONDARY OUTCOMES:
Changes in fasting blood glucose response in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  fasting blood glucose response in 12-week intervention
Changes in fasting blood insulin response in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  fasting blood insulin response in 12-week intervention
Changes in fasting HbA1c response in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  fasting HbA1c response in 12-week intervention
Changes in blood pressure in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  blood pressure in 12-week intervention
Changes in fasting blood Triglycerides concentration in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  fasting blood Triglycerides concentration in 12-week intervention
Changes in fasting hs C-Reactive Protein in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  fasting hs C-Reactive Protein in 12-week intervention
Changes in fasting markers of endothelial dysfunction (ICAM-1) in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  fasting markers of endothelial dysfunction (ICAM-1) in 12-week intervention
Changes in fasting markers of endothelial dysfunction (VCAM-1) in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  fasting markers of endothelial dysfunction (VCAM-1) in 12-week intervention
Changes in attitudes towards eating measured by the Stunkard 3-Factor Eating Questionnaire in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  attitudes towards eating measured by the Stunkard 3-Factor Eating Questionnaire in 12-week intervention
Changes in plasma LDL cholesterol in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  plasma LDL cholesterol in 12-week intervention
Changes in plasma total cholesterol in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  plasma total cholesterol in 12-week intervention
Changes in plasma HDL cholesterol in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  plasma HDL cholesterol in 12-week intervention

OTHER OUTCOMES:
Changes in body weight in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  body weight in 12-week intervention
Changes in waist circumference in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  waist circumference in 12-week intervention
Changes in body composition in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  body composition in 12-week intervention
Changes in blood lipoproteins in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  Changes in lipoprotein particle size/density by nuclear magnetic resonance (NMR)
Changes in blood IL-6 in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  blood IL-6 in 12-week intervention
Changes in blood MCP-1 in 12-week intervention of active treatment vs control treatment. | baseline and 12 weeks
  blood MCP-1 in 12-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Britt Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Xiao D, Guzman G, Edirisinghe I, Burton-Freeman B. Avocado Consumption for 12 Weeks and Cardiometabolic Risk Factors: A Randomized Controlled Trial in Adults with Overweight or Obesity and Insulin Resistance. J Nutr. 2022 Aug 9;152(8):1851-1861. doi: 10.1093/jn/nxac126. PMID 35700149